CLINICAL TRIAL: NCT05792111
Title: Analgesic Effects of Trigger Point Injection Added to Caudal Epidural Steroid
Brief Title: Caudal Epidural Steroid and Trigger Point Injection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Murat Bilgi, Prof.dr, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AİBU-Med-MB-01
Record Dates: First submitted 2022-10-18; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Myofascial Trigger Point Pain
Keywords: Caudal Epidural Steroid Injection; Trigger Point Injection; NRS score
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Lidocaine; Bupivacaine; Triamcinolone

STUDY DESIGN:
Intervention Model Description: Trigger point injection was added to the gluteus medius and gluteus Maximus muscles in addition to caudal epidural steroids.
Who Masked: Investigator
Masking Description: The staff who will evaluate the patient before and after the procedure will not know which group the patients belong to, and the study will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Experimental): Group C; caudal epidural steroid injection (10 mL volume of bupivacaine 4cc/20mg+ triamcinolone 2cc/80mg+0.09% NaCl 4cc mixture will be administered into the caudal epidural space).
  Interventions: Drug: Caudal epidural Group (bupivacaine + triamcinolone + NaCl)
- Group CT (Active Comparator): Group CT; trigger point injection will be added to the gluteus medius and minimus muscles in addition to caudal epidural steroid injection.
  Interventions: Drug: Trigger point injection (lidocaine); Drug: Caudal epidural Group (bupivacaine + triamcinolone + NaCl)

INTERVENTIONS:
Drug: Trigger point injection (lidocaine) — trigger point injection will be added to the gluteus medius and minimus muscles in addition to caudal epidural steroid injection.
  Other Names: lidocaine
  Arms: Group CT
Drug: Caudal epidural Group (bupivacaine + triamcinolone + NaCl) — It will be advanced towards the sacral hiatus and local anesthesia of the skin and subcutaneous tissue will be provided with 2% lidocaine. The caudal epidural space will be entered by puncturing the sacrococcygeal ligament with the tip of a 22 G black needle from the appropriate area and taking a pop sensation. It will be confirmed that there is no bleeding or cerebrospinal fluid in this area by applying saline in real-time sonography and after the caudal epidural spread is observed, aspiration is performed. Afterward, a 10 mL volume of bupivacaine 4cc/20mg+ triamcinolone 2cc/80mg+0.09% NaCl 4cc mixture will be administered into the caudal epidural space
  Other Names: triamsinolon asetonid

SUMMARY:
This prospective randomized study will be conducted in Bolu Abant İzzet Baysal University Hospital. Chronic low back and hip pain 72 patients aged between 18-70 years will be included in the study. The primary output of our study was NRS scores. The study of Manchikanti. L et al. (control group NRS reduction 4.4 ± 1.8; α margin of error 0.05, power 99%) (3) was taken as the basis for determining the sample size. Using the G Power 3 calculator program, 72 patients were identified to reduce their NRS scores by 25%. With a 20% exclusion rate, the total number of patients was calculated as 90

DETAILED DESCRIPTION:
Demographic information of all patients included in the study; name, surname, telephone number, age, gender, educational status, profession, and marital status will be recorded. The duration of the pain, the onset of the pain, the accompanying leg pain, the activities that increase or decrease the pain, the presence of neurological symptoms, the analgesic agents used in the last week, and the previous treatments will be noted. Lumbar MRI findings and the level of pathology causing low back and hip pain will be recorded. History, family history, comorbidities (hypertension, diabetes mellitus, hyperlipidemia, cardiac disease, hypothyroidism), and detailed physical examinations of the patients will be recorded. Examinations of the patients before and 3, 6, and 12 weeks after the injection will be performed, and NRS scores at 3 and 6 weeks. The procedures will be repeated for patients who are over 4 years old. During the pre-procedural evaluation, the patients will be informed about the study, information about the Numeric Rating Score (NRS), Oswestry Disability Index (ODI), Short Form-36 (SF-36) to be used for post-procedure analgesia, and both verbal and written consents will be obtained. The staff who will make the evaluation will not know which group the patients belong to, and the study will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Low back or leg pain that has been going on for at least 2 months,
* Patients between the ages of 18-70,
* Disc herniation or radiculopathy in lumbar MRI examination .To be mentally competent to understand and evaluate NRS, ODI, and SF-36 forms.

exclusion criteria

* Being pregnant or lactating,
* Presence of spinal canal stenosis,
* The presence of bleeding diathesis,
* Presence of disease with progressive neurological deficit,
* The presence of serious psychiatric illness,
* Presence of progressive neurological deficit or incontinence,
* Having an epidural steroid injection in the last 6 months, Having uncontrolled diabetes mellitus Having hypertension,
* Known history of allergy to local anesthetics or corticosteroids,
* The patient does not want treatment,
* Local infection at the injection site,
* Infections such as discitis, spondylodiscitis, and sacroiliitis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) score | basaline,
  NRS score measures a patient's pain intensity. For example, (range 0-10) where 0 is no pain and 10 is the worst pain
Numerical Rating Scale (NRS) score | after ESİ 3 weeks,
  NRS score measures a patient's pain intensity. For example, (range 0-10) where 0 is no pain and 10 is the worst pain
Numerical Rating Scale (NRS) score | after ESİ 6 weeks
  NRS score measures a patient's pain intensity. For example, (range 0-10) where 0 is no pain and 10 is the worst pain
Numerical Rating Scale (NRS) score | after ESİ12 weeks
  NRS score measures a patient's pain intensity. For example, (range 0-10) where 0 is no pain and 10 is the worst pain

SECONDARY OUTCOMES:
Oswestry Disability Index | basaline
  used to qualify low back pain.(range 0 to 100).Zero is equated with no disability and 100 is the maximum disability possible
Oswestry Disability Index | after ESİ 3 weeks
  used to qualify low back pain.(range 0 to 100).Zero is equated with no disability and 100 is the maximum disability possible
Oswestry Disability Index | after ESİ 6 weeks
  used to qualify low back pain.(range 0 to 100).Zero is equated with no disability and 100 is the maximum disability possible
Oswestry Disability Index | after ESİ12 weeks
  used to qualify low back pain.(range 0 to 100).Zero is equated with no disability and 100 is the maximum disability possible
Short Form-36 | basaline
  used to measure of patient's health status.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Short Form-36 | after ESİ 3 weeks,
  used to measure of patient's health status.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Short Form-36 | ,after ESİ 6 weeks
  used to measure of patient's health status.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Short Form-36 | after ESİ12 weeks
  used to measure of patient's health status.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University Medical School,, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No